CLINICAL TRIAL: NCT04470310
Title: Comparison of Glimepiride, Alogliptin and Alogliptin+Pioglitazone Combination in Poorly Controlled Type 2 Diabetic Patients
Brief Title: Glimepiride, Alogliptin and Alogliptin+Pioglitazone Combination
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung Hee Choi, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Takeda_ALO-IIT
Record Dates: First submitted 2020-07-01; First posted 2020-07-14 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; alogliptin

STUDY DESIGN:
Intervention Model Description: Group A (glimepiride), Group B (alogliptin), and Group C (alogliptin-pioglitazone)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- glimepiride (Active Comparator): glimepiride 1mg monotherapy and glimepiride 2mg monotherapy
  Interventions: Drug: Glimepiride
- alogliptin (Active Comparator): alogliptin 25mg monotherapy
  Interventions: Drug: Alogliptin 25Mg Tab
- alogliptin - pioglitazone (Active Comparator): Alogliptin 25mg+pioglitazone 15mg combination
  Interventions: Drug: Alogliptin-Pioglitazone 25 Mg-15 Mg Oral Tablet

INTERVENTIONS:
Drug: Glimepiride
  Arms: glimepiride
Drug: Alogliptin 25Mg Tab
  Arms: alogliptin
Drug: Alogliptin-Pioglitazone 25 Mg-15 Mg Oral Tablet
  Arms: alogliptin - pioglitazone

SUMMARY:
* This trial is a three-armed, open label, random assignment trial.
* The research subjects are patients who are first starting their treatment or patients who have failed with the metformin treatment and are changing their medication. They will be assigned to one of the following treatment groups: the glimepiride monotherapy treatment group, the alogliptin monotherapy treatment group, and the alogliptin - pioglitazone combination therapy treatment group
* This trial is a prospective trial which will conduct surveys 6 times over the course of the 6 months in which each treatment group is administered drugs (Week -2, Baseline, Week 4, Week 12, Week 24, follow-up safety survey).
* This trial is a multicenter clinical trial which will be conducted at more than 5 general hospital medical institutions in the vicinity of the capital.

DETAILED DESCRIPTION:
* The research subjects selected for this trial will patients among those who have given their approval to participate in the trial and who are first starting their treatment or who intend to alter their medication because treatment with the existing drugs has failed who satisfy the criteria.
* Patients with a '7.5% ≤ HbA1c ≤ 10%' in the HbA1c test will be chosen.
* Patients who are intending to change drugs due to the failure of an existing drug treatment must have the use of 1,000 mg or the maximum tolerance dose (MTD) of metformin recorded in his or her medical records.
* The investigators must confirm the patient's intention to participate in the trial and, starting at the point of the routine laboratory test results, must provide a sufficient explanation of this research to the patients who satisfy the criteria and then must acquire a research subject consent form from these patients. The consent forms must include the trial objectives, the benefits for participants, the risk factors, a confidentiality agreement, the right to withdraw consent, and contact information. The patients must sign the consent forms.

  * The change in the level of HbAc1 will be compared among the 3 treatment groups - the glimepiride monotherapy treatment group, the alogliptin monotherapy treatment group, and the alogliptin - pioglitazone combination therapy treatment group - until the 24th week after the Baseline is taken.
  * CGMS will be checked to investigate changes in blood glucose.
  * Glimepiride's nonproprietary name is glimepiride; this drug is a snowman shaped tablet. Starting with a 1 mg dosage once a day before the first meal, the investigators will decide to increase the dosage to a maximum of 2 mg in the Week 4.
  * Dosage adjustment will be conducted for participants proven to have persistent hyperglycemia (in the opinion of the investigator).

Week 4 Week 12 Alogliptin 25mg Dosage adjustment is not allowed Dosage adjustment is not allowed Glimepiride1mg 2mg Dosage adjustment is not allowed Alogliptin 25mg

+Pioglitazone 15mg Dosage adjustment is not allowed Dosage adjustment is not allowed

* Alogliptin's nonproprietary name is alogliptin benzoate and is an oval-shaped yellow tablet. A 25 mg dose of this medication is administered once a day and is taken with food or on an empty stomach.
* The pioglitazone used by the alogliptin - pioglitazone combination therapy treatment group is pioglitazone hydrochloride and is a grey circular tablet. A 15 mg dose of this medication is administered once a day and is taken with food or on an empty stomach.
* The subjects will test the HbA1c level in Week 12 and Week 24 and will check CGMS at the Baseline and in Week 24.
* General characteristics (bodyweight and BMI), vital signs, and laboratory tests will be conducted in Week 4, Week 12, and Week 24.
* MAGE will be measured using CGMS (continuous glucose monitoring system) for 3 days (72 hours). Education regarding eating, CGMS usage, notices, and correction will be given.
* A follow-up safety survey will be conducted 30 days after the last visit.
* Subjects will be enrolled in the trial for 6 months and following this a follow-up survey will be conducted.
* Approximately 12 months will be required for the total trial period based on the last patient (6 months) to have their Baseline enrollment conducted.
* Patients will be asked to come to the clinical research institution after Week 4, Week 12, and Week 24 (for Week 12 and Week 24, a period of ±7 days is permitted) after the Baseline (or the first) visit. In addition, patients will be requested to take a call 30 days after their last visit for the safety follow-up survey.
* Subjects with a drug compliance of less than 80% will be eliminated.
* Subjects with an HbA1c level of more than 9.0% in Week 12 will be eliminated. Subjects who sign the trial subject consent form and participate in the trial but do not finish will be eliminated. The elimination of a subject can be determined at any time during the trial. Withdrawal of consent by the subject will also be considered as an elimination and the reason for the withdrawal of consent must be clearly recorded. Furthermore, if an adverse event and/or a serious adverse event occurs during the trial, the corresponding subject will be immediately eliminated from the trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects selected for this trial will be male and female outpatients 19 - 80 years of age (by date of birth) with type 2 diabetes and with HbA1c levels of 7.5%≤HbA1c≤10%.
* Patient's body mass index must be greater than 18 kg/m2.
* Subjects selected for the trial are patients who are starting treatment for the first time or who have failed with more than 8 weeks of treatment with 1,000 mg or the maximum tolerance dose (MTD) of metformin and want to change their medication.

Exclusion Criteria:

* If weight loss pills were used in the last 3 months, or hypoglycemic agents or lipid lowering agents used in a clinical trial (not including statins or ezetimibe) were used in the last 3 months.
* If the subject received systemic corticosteroid treatment or there was a change in the dosage of thyroid hormones in the 6 weeks prior to the study.
* If insulin was used within the 3 months prior to screening.
* If the patient's C-peptide level is less than 0.6 ng/mL.
* If an allergy or a hypersensitivity reaction to the target drug or its ingredients occurs.

Additional criteria for exclusion are listed below;

* A medical history of type 1 diabetes; acute metabolic complications of diabetes within the past 6 months (e.g., ketoacidosis or a hyperosmolar state (coma or precoma))
* Hematological disorder
* A medical history of angioedema caused by angiotensin converting enzyme inhibitors or angiotensin receptor blockers or a medical history of treatment for diabetic gastroparesis
* If there are clear symptoms of hypothyroidism or hyperthyroidism in the opinion of the investigator.
* Myocardial infarction or percutaneous coronary intervention (stent nephrostomy or balloon nephrostomy) within the past 6 months
* Serious heart failure or a medical history of heart failure (NYHA Class III or IV heart failure)
* Heart failure, moderate to severe kidney injury (creatinine clearance of <50 mL/min prior to screening)
* Patients with chronic hepatitis, or hepatitis B or C (not including healthy carriers of hepatitis B) or a patient with liver disease (defined as cases in which the alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, or serum total bilirubin level is higher than 2.5 times the ULN)
* Hereditary complications, such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption (restricted to drugs including lactase)
* Cardiovascular disease or myocardial infarction; or a percutaneous transluminal coronary angioplasty or coronary artery stent nephrostomy within the past 6 months
* A serious cerebrovascular accident, stroke, or transient ischemic attack within the past 6 months
* Laser treatment for diabetic proliferative retinopathy
* A medical history of alcohol or drug abuse in the past 3 months
* A medical history of cancer in which remission could not be achieved within 5 years
* A medical history of bladder cancer or active bladder cancer
* Uninvestigated macroscopic hematuria
* Has experienced major surgery
* Breast feeding women, pregnant women, or premenopausal for whom pregnancy is possible are not suitable for participation in this trial
* External injury, acute infection, existence of or medical history of other chronic illness

Criteria for exclusion based on laboratory test results are as listed below.

* A fasting blood glucose (FPG) level of >239.6 mg/dL
* Systolic or diastolic blood pressure of >160 mmHg or >100 mmHg respectively
* A serum creatinine level of 1.5 mg/dL for men or 1.4 mg/dL for women
* An albumin/creatinine ratio of 2,000 mg/g
* A fasting triglyceride level of > 5.1 mmol/l (452 mg/dL)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline, Week 24
  The change in the mean level of HbA1c from baseline at week 24

SECONDARY OUTCOMES:
HbA1c and fasting plasma glucose | Baseline, Week 12, Week 24
  The change in the mean level of HbA1c at week 12 and mean FPG( fasting plasma glucose) levels
The change in parameters of glycemic variability assessed by CGM from the Baseline at week 24 | Baseline, Week 24
  The change in parameters of glycemic variability assessed by CGM from baseline at week 24: SD(standard deviation), MAGE(Mean Amplitude of Glycaemic Excursions); MODD(Mean of Daily Differences); ADDR(Average Daily Risk Range), M-value
The change in lipid profile from baseline at week 12 and 24 | Baseline, Week 12, Week 24
  The average change in the lipid profile: Total cholesterol (mg/dL), Triglyceride(mg/dL), HDL-cholesterol, (mg/dL) LDL cholesterol (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Hee Choi, Principal Investigator — Seoul National University Hospital

DOCUMENTS (1):
  • Study Protocol (2016-12-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT04470310/Prot_000.pdf